CLINICAL TRIAL: NCT00232284
Title: An Integrated Pharmacological and Psychological Approach to Young People With Comorbid Depression and Substance Abuse
Brief Title: Treatment of Comorbid Depression and Substance Abuse in Young People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Lubman (Other)
Responsible Party: Sponsor-Investigator, Dan Lubman, Dr Dan Lubman, Melbourne Health
Organization: Melbourne Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MHREC 2004.030
Record Dates: First submitted 2005-10-02; First posted 2005-10-04 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Depression; Substance-Related Disorders
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertaline (Active Comparator): 8 week course of sertraline 50-100mg for those who fail to respond to CBT within first 4 weeks of study entry
  Interventions: Drug: sertraline; Behavioral: Cognitive Behavioural Therapy
- Placebo (Placebo Comparator): 8 week course of placebo
  Interventions: Drug: sertraline; Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Drug: sertraline — RCT of sertraline/placebo for those young people who fail to respond within first 4 weeks of study entry
  Other Names: Zoloft
Behavioral: Cognitive Behavioural Therapy — An integrated 10-week CBT program for depression/anxiety and comorbid substance use
  Other Names: CBT

SUMMARY:
This study aims to treat young people with an adjunctive integrated cognitive behavioral therapy (CBT) intervention and to examine the acceptability of this treatment approach within this population. The study will also include a pilot placebo-controlled trial of sertraline for those young people who fail to or only partially respond to the CBT intervention, so as to determine whether adjunctive anti-depressant treatment improves clinical response in this population.

DETAILED DESCRIPTION:
The high prevalence of co-occurring depressive and substance use disorders amongst young people is especially problematic given the significant negative impact on both symptom course and outcome reported in adult samples. Whilst the clinical and functional outcomes in young people with comorbid disorders remains largely unknown, of particular concern is the consistent association between depression, substance misuse and suicidality in young people, especially given the high rates of youth suicide in Australia. As such, it is both a clinical priority and an important public health goal that the clinical characteristics and outcomes of young people with comorbid depression and substance abuse are identified, and that effective biopsychosocial interventions are developed that encompass predictors of treatment, such that targeted integrated treatments may be offered wherever affected young people present.

Whilst there is strong evidence for both selective serotonin reuptake inhibitors (SSRIs) and CBT in the treatment of depression, and some support for their utility in alcohol dependence, no studies have examined their utility in a group of young people with comorbid depression and substance abuse. In fact, whilst CBT is suggested to be the first-line treatment for depression in young people, its role in comorbid disorders is less clear, and there is little data on predictors of treatment outcome in this population. Which young people best respond and which do not are important questions when designing the most appropriate interventions for real-world clinical settings. In this regard, the role of anti-depressants in comorbid populations also remains contentious, especially amongst those that fail or only partially respond to CBT. In particular, it is unclear at what stage anti-depressants should be offered or even whether SSRIs are indeed effective in this population.

Research Questions This project encompasses two complementary studies that aim to examine the characteristics and outcomes of young people with comorbid depression and substance abuse. Stage 1 is a preliminary naturalistic investigation of the characteristics of young people with comorbid depressive and substance use disorders presenting to drug treatment and mental health services, and describes their outcomes over 6, 12 and 24 months. This study seeks to explore what happens to these young people in the current service system, in terms of engagement and treatment, and related substance use and mental health outcomes. Stage 2 aims to treat a sub-sample of these young people with an adjunctive integrated CBT intervention and to examine the acceptability of this treatment approach within this population. In addition, this study seeks to explore predictors of treatment outcome so as to inform the further development of this integrated intervention. Stage 2 will also include a pilot placebo-controlled trial of sertraline for those young people who fail to or only partially respond to the CBT intervention, so as to determine whether adjunctive anti-depressant treatment improves clinical response in this population.

The specific aims of the study are:

* To describe the course of depressive disorders amongst young people with comorbid substance use disorders
* To explore predictors of treatment response to an integrated CBT intervention
* To explore the acceptability of the CBT intervention within a comorbid youth population
* To explore the role of sertraline in the treatment of non-response to CBT in a comorbid youth population

ELIGIBILITY:
Inclusion Criteria:

* 16 and 26 years of age
* acute major depressive episode (more than one month)
* concurrent DSM-IV substance abuse/dependence or the use of any illicit drug on a weekly basis in the month prior to referral, or alcohol consumption exceeding NHMRC guidelines
* English as their preferred language
* estimated IQ >80

Exclusion Criteria:

* Current or past history of psychosis
* significant head injury
* seizures
* history or current evidence of any other significant clinical condition
* treatment with an antidepressant within past 30 days

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2004-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
HAMD depression at 10 weeks, 20 weeks and 44 weeks | 10 weeks, 20 weeks and 44 weeks
OTI TLFB substance use levels at same time points | 10 weeks, 20 weeks and 44 weeks

SECONDARY OUTCOMES:
MASQ self report mood and anxiety at 10 weeks, 20 weeks and 44 weeks | 10 weeks, 20 weeks and 44 weeks
DAS self report dysfunctional attitudes at same time points | 10 weeks, 20 weeks and 44 weeks
ATQ self report automatic thoughts at same time points | 10 weeks, 20 weeks and 44 weeks
SDS self report severity of dependence at same time points | 10 weeks, 20 weeks and 44 weeks
DUMM self report drug use motives at same time points | 10 weeks, 20 weeks and 44 weeks
RTC self report readiness to change at same time points | 10 weeks, 20 weeks and 44 weeks
CISS self report coping with stress at same time points | 10 weeks, 20 weeks and 44 weeks
CGI severity of illness at same time points | 10 weeks, 20 weeks and 44 weeks
SOFAS social and occupational functioning at same time points | 10 weeks, 20 weeks and 44 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lubman, Principal Investigator — ORYGEN Youth Health, University of Melbourne, Department of Psychiatry
Locations (1):
- ORYGEN Youth Health, Melbourne, Victoria, Australia